CLINICAL TRIAL: NCT01159548
Title: Efficacy of Low Dose Promethazine for Postoperative Nausea and Vomiting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Population of interest was no longer available
Sponsor: Women's College Hospital (Other)
Responsible Party: Dr. Jean Kronberg, Women's College Hospital
Allocation: Randomized | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-0034B
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Ambulatory Gynecological Laparoscopic Procedures
MeSH Terms: interventions — Promethazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline (No Intervention)
- Promethazine 6.25 mg (Other)
  Interventions: Drug: Promethazine
- Promethazine 3 mg (Other)
  Interventions: Drug: Promethazine

INTERVENTIONS:
Drug: Promethazine
  Arms: Promethazine 6.25 mg
Drug: Promethazine
  Arms: Promethazine 3 mg

SUMMARY:
There has been an increase in ambulatory surgical procedures performed across Canada; ambulatory procedures account for almost 70% of all surgeries. Postoperative nausea and vomiting (PONV) and pain are the most frequently reported adverse events by patients prior to discharge after ambulatory surgery. The incidence can be as high as 70 to 80% in high-risk patients.

PONV is a cause of morbidity particularly in gynecological procedures and the incidence of patients experiencing PONV is as high as 58-75%. Apart from delayed recovery, the occurrence of PONV has been linked to gastric aspiration, psychological distress and wound dehiscence. The occurrence of PONV delays patient discharge and further more is a leading cause of unexpected admission after ambulatory anesthesia

Promethazine, is an antiemetic medication that has been widely used over the last 50 years, and although effective at reducing PONV, it tends to cause sedation. In this study, we are trying to determine if a smaller dose of promethazine, in addition to the standard treatment for post-surgical nausea and vomiting, will be more beneficial than the standard treatment on its own.

It is hypothesized that the use of low dose promethazine (3 mg) as part of a multimodal antiemetic regimen will be efficacious in preventing PONV without the sedative effects of promethazine.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 - 60 yrs of age

2 Patient's health is graded as class I-III according to the American Society of Anesthesiologists physical status classification.

3. The patient has 2 or more of the following risk factors:

* Female
* Non-smoker
* History of PONV/motion sickness
* Use of post-operative opioids (current surgery)

  4. Undergoing ambulatory gynecological laparoscopic procedures of at least 30 minutes duration

Exclusion Criteria:

* preexisting nausea, vomiting or retching, gastric outlet or intestinal obstruction
* clinical evidence of a difficult airway
* obesity (body mass index > 40 kg m-2)
* scheduled to receive propofol for anesthesia maintenance
* current pregnancy
* psychiatric illness
* clinically significant major organic disease
* preoperative QTc interval > 440 ms on electrocardiogram
* known hypersensitivity to promethazine, granisetron, ondansetron or other 5 HT3-receptor antagonists

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Absence of emetic episode for 24 h in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Jean Kronberg, MD, PhD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada